CLINICAL TRIAL: NCT02182830
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group, Efficacy and Safety Study of Empagliflozin (10mg, 25mg) Administered Orally, Once Daily Over 24 Weeks in Hypertensive Black/African American Patients With Type 2 Diabetes Mellitus
Brief Title: 24 Week Efficacy and Safety Study of Empagliflozin (BI 10773) in Hypertensive Black/African American Patients With Type 2 Diabetes Mellitus and Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.29
Record Dates: First submitted 2014-07-03; First posted 2014-07-08 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — empagliflozin

ARMS (2):
- Empagliflozin (Experimental): starting dose 10mg; forced titration after 4 weeks 25mg dose
  Interventions: Drug: Empagliflozin low dose; Drug: Empagliflozin high dose
- Placebo (Placebo Comparator): starting dose 10mg; forced titration after 4 weeks 25mg dose
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Empagliflozin low dose — starting dose 10mg; forced titration after 4 weeks 25mg dose
  Arms: Empagliflozin
Drug: placebo — starting dose 10mg; forced titration after 4 weeks 25mg dose
  Arms: Placebo
Drug: Empagliflozin high dose — starting dose 10mg; forced titration after 4 weeks 25mg dose
  Arms: Empagliflozin

SUMMARY:
This trial is designed to investigate the efficacy and safety of empagliflozin compared with placebo in hypertensive black/African Americans with type 2 Diabetes Mellitus. Since hyperglycaemia and hypertension are key risk factors for both micro- and macrovascular complications, assessment of both glucose and BP lowering effects of empagliflozin in hypertensive African American patients with type 2 Diabetes Mellitus could provide clinically highly relevant, new information for the use of empagliflozin.

Essential hypertension is four times more common in African Americans than in Caucasians.

One of the risk factors for hypertension is sodium sensitivity and approximately one third of the essential hypertensive population is responsive to sodium intake. There is a higher association of hypertension with sodium sensitivity in African American patients with type 2 Diabetes Mellitus.

The treatment duration of this trial (24 weeks) will enable assessment of the clinically relevant endpoint of a decrease in HbA1c, a well accepted measurement of chronic glycaemic control and the key secondary endpoints of decreases in systolic BP (SBP) and diastolic BP (DBP) at 12 and 24 weeks.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of Type 2 Diabetes Mellitus (T2DM) prior to informed consent.
* Male and female black/African American patients on diet and exercise regimen who are EITHER drug-naïve (defined as absence of any oral antidiabetic therapy, glucagon like peptide-1 (GLP-1) analog or insulin for 12 weeks, 16 weeks for pioglitazone prior to randomisation) OR pre-treated with stable dose of

  * Metformin only, or
  * Sulfonylurea only, or
  * Dipeptidyl peptidase-4 (DPP-4) inhibitor only, or
  * metformin plus sulfonylurea, or
  * metformin plus DPP-4 inhibitor. Treatment has to be unchanged for a minimum of 12 weeks prior to randomization. Dose for metformin: maximum tolerated dose The maximum daily dose of Sulfonylurea (SU) or DPP-4 inhibitor should not exceed that stated in the local label.
* HbA1c of >= 7.0% (53 mmol/mol) and ≤ 11.0% (97 mmol/mol) at Visit 1 (screening).
* Mean seated Systolic Blood Pressure (SBP) 140-180 mmHg at Visit 1 (screening).
* Successful completion of baseline Ambulatory Blood Pressure Monitor (ABPM) testing with a mean SBP 135-175 mmHg prior to randomisation.
* Treatment with stable doses of at least one but not more than 4 antihypertensive medication >= 4 weeks prior to randomisation.
* Age >= 18 years at Visit 1 (screening)
* Signed and dated written informed consent by date of Visit 1 in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

* Uncontrolled hyperglycemia with a glucose level >270 mg/dl (>15.0 mmol/L) after an overnight fast during placebo run-in (includes Visit 2.1) and confirmed by a second measurement (not on the same day).
* Exposure to any other antidiabetic medication within 12 weeks prior to randomisation other than metformin, sulfonylurea, Dipeptidyl peptidase-4 (DPP-4) inhibitor, metformin plus sulfonylurea or metformin plus DPP-4 inhibitor.
* Current hypertension treatment with oral Minoxidil (topical minoxidil for hair growth is allowed).
* Mean seated Systolic Blood Pressure (SBP) ≥181 mmHg during placebo run-in visit and confirmed by a second measurement (not on the same day) preferably within one day.
* Upper arm circumference that exceeds the upper circumference level of the cuff size of either Ambulatory Blood Pressure Monitor (ABPM) and/or (BP) measurement device used in the study.
* Night shift workers who routinely sleep during the daytime and/or whose work hours include midnight.
* Diagnosis of autoimmune diabetes/Type I diabetes mellitus, monogenic (neonatal or maturity onset diabetes of the young (MODY)) diabetes or Type I diabetes in adults/latent autoimmune diabetes of adults (LADA) per investigator or patient medical history at the time of Visit 1 (screening).
* Known or suspected secondary hypertension (e.g. renal artery stenosis,phaeochromocytoma, Cushing's disease).
* History or evidence of hypertensive retinopathy (Keith-Wagener grade III or IV) and/or hypertensive encephalopathy.
* Clinically significant valvular heart disease or severe aortic stenosis in the opinion of the investigator.
* Acute coronary syndrome (non- ST wave elevated myocardial infarction (STEMI), STEMI and unstable angina pectoris), stroke or transient ischemic attack within 3 months prior to informed consent.
* Indication of liver disease, defined by serum levels of either Alanine Aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase(SGPT)), Aspartate Aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)), or alkaline phosphatase above 3 x upper limit of normal (ULN) as determined during screening and/or run-in phase.
* Impaired renal function, defined as Estimated Glomerular Filtration Rate (eGFR)< 45 ml/min/1.73m2 (moderate renal impairment, chronic kidney disease epidemiology collaboration Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula) as determined during screening and/or run-in phase.
* Bariatric surgery within the past two years and other gastrointestinal surgeries that induce chronic malabsorption.
* Medical history of cancer (except for basal cell carcinoma) and/or treatment for cancer within the last 5 years.
* Blood dyscrasias or any disorders causing hemolysis or unstable Red Blood Cells (e.g. malaria, babesiosis, haemolytic anaemia, thalassemia, sickle cell anaemia (sickle cell trait is allowed)).
* Medical history and signs and symptoms of diabetic autonomic neuropathy.
* Treatment with anti-obesity drugs 3 months prior to randomisation (i.e. surgery, aggressive diet regimen, etc.) leading to unstable body weight.
* Current treatment with systemic steroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent or any other uncontrolled endocrine disorder except Type 2 Diabetes Mellitus (T2DM) in the opinion of the investigator.
* Pre-menopausal women (last menstruation <=1 year prior to informed consent) who:

  * are nursing or pregnant or
  * are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial. Acceptable methods of birth control include tubal ligation, transdermal patch, intra uterine devices/systems (IUDs/IUSs), oral, implantable or injectable contraceptives, complete sexual abstinence (if acceptable by local authorities), double barrier method and vasectomised partner.
* Alcohol, drug or confectionary liquorice abuse within the 3 months prior to informed consent that would interfere with trial participation or any ongoing condition leading to a decreased compliance to study procedures or study drug intake in the investigator's opinion.
* Intake of an investigational drug in another trial within 30 days prior to intake of study medication in this trial; or participating in another trial (involving an investigational drug and/or follow-up) after discontinuing medication in that trial.
* Any other clinical condition that would jeopardize patient's safety while participating in this clinical trial in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2014-07-25 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2017-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (92):
- United States (92):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Clinical Research Advantage, Inc./Rita B. Chuang, MD, LLC, Birmingham, Alabama
  - Longwood Research, Huntsville, Alabama
  - Internal Medicine Center, LLC, Mobile, Alabama
  - Mobile Medical and Diagnostic Center, Mobile, Alabama
  - University of South Alabama, Mobile, Alabama
  - Cardiology and Medicine Clinic, Little Rock, Arkansas
  - Larry Watkins, M .D., Little Rock, Arkansas
  - eStudySite, Chula Vista, California
  - Torrance Clinical Research Institute Inc., Lomita, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - MD Clinical Trials, Los Angeles, California
  - Office of Dr. Alexander Ford, M.D., Los Angeles, California
  - Diabetes Associates Medical Group, Orange, California
  - Integrated Research Group, Inc., Riverside, California
  - Clinical Trials Research, Sacramento, California
  - Orange County Research Center, Tustin, California
  - Lynn Institute of Denver, Denver, Colorado
  - Pines Clinical Research Inc., Hollywood, Florida
  - UF Health Jacksonville, Jacksonville, Florida
  - Care Partners Clinical Research LLC, Jacksonville, Florida
  - Sunshine Research Center, Opa-locka, Florida
  - Central Florida Internist, Orlando, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - International Clinical Research - US, LLC, Sanford, Florida
  - Meridien Research, St. Petersburg, Florida
  - Alternative Solutions Medical Research and Prevention Center, St. Petersburg, Florida
  - Meridien Research, Tampa, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Morehouse School of Medicine, Atlanta, Georgia
  - Atlanta Center, Atlanta, Georgia
  - Atlanta Clinical Research Centers, Atlanta, Georgia
  - Albert F. Johary MD, PC, Dunwoody, Georgia
  - Sestron Clinical Research, Marietta, Georgia
  - Clinical Research Advantage, Inc./Rita B. Chuang, MD, LLC, Marietta, Georgia
  - WR-Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Eagle's Landing Diabetes and Endocrinology, Stockbridge, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - John H. Stroger Jr. Hospital of Cook Country, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Investigators Research Group, LLC, Brownsburg, Indiana
  - Centex Studies, Inc., Lake Charles, Louisiana
  - Gulf Regional Research and Education Services, LLC, Metairie, Louisiana
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - American Institute of Research Studies, Baltimore, Maryland
  - Phillips Medical Services, PLLC, Jackson, Mississippi
  - Mercy Research, Washington, Missouri
  - Quality Clinical Research Inc, Omaha, Nebraska
  - Accent Clinical Trials, Las Vegas, Nevada
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - Offic of Dr. Eric Cheng, Brooklyn, New York
  - Healthwise Medical Associates, Brooklyn, New York
  - Modern Medical, Brooklyn, New York
  - Erie County Medical Center, Buffalo, New York
  - Scott Research, Inc., Laurelton, New York
  - Medex Healthcare Research, Inc., New York, New York
  - Laurelton Heart Specialist, PC, Rosedale, New York
  - Metrolina Internal Medicine, PA, Charlotte, North Carolina
  - PhysiqueMed Clinical Trials, Greensboro, North Carolina
  - Triad Clinical Trials, Greensboro, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - High Point Clinical Trials Center, High Point, North Carolina
  - Coastal Carolina Health Care, P.A., New Bern, North Carolina
  - Hometown Urgent Care, Columbus, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - Today Clinical Research, Oklahoma City, Oklahoma City, Oklahoma
  - Suburban Research Associates, Media, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Medical Research South, Charleston, South Carolina
  - TLM Medical Services, LLC, Columbia, South Carolina
  - Amistad Clinical Research Center, Columbia, South Carolina
  - Greenville Pharmaceutical Rsch, Greenville, South Carolina
  - Mountain View Clinical Research, Greer, South Carolina
  - Berkley Family Practice, Moncks Corner, South Carolina
  - Carolina Cardiology Clinical Research Institute, LLC, Rock Hill, South Carolina
  - Community Research Partners, Inc, Varnville, South Carolina
  - Memphis Veterans Affairs Medical Center, Memphis, Tennessee
  - The Green Clinic PC, Memphis, Tennessee
  - Southwind Medical Specialists, Memphis, Tennessee
  - University of Tennessee, Memphis, Tennessee
  - Diagnostic Clinic of Houston, Houston, Texas
  - Cullen Family Practice, PLLC, Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Kelsey-Seybold Clinic, Houston, Texas
  - Hillcrest Family Health Center, Waco, Texas
  - Millennium Clinical Trials LLC, Arlington, Virginia
  - York Clinical Research, LLC, Norfolk, Virginia
  - Dominion Medical Associates, Inc., Richmond, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Family Medical Clinic, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Ferdinand KC, Harrison D, Johnson A. The NEW-HOPE study and emerging therapies for difficult-to-control and resistant hypertension. Prog Cardiovasc Dis. 2020 Jan-Feb;63(1):64-73. doi: 10.1016/j.pcad.2019.12.008. Epub 2020 Jan 8. PMID 31923435
- [Derived] Ferdinand KC, Izzo JL, Lee J, Meng L, George J, Salsali A, Seman L. Antihyperglycemic and Blood Pressure Effects of Empagliflozin in Black Patients With Type 2 Diabetes Mellitus and Hypertension. Circulation. 2019 Apr 30;139(18):2098-2109. doi: 10.1161/CIRCULATIONAHA.118.036568. PMID 30786754
- [Derived] Ferdinand KC, Seman L, Salsali A. Design of a 24-week trial of empagliflozin once daily in hypertensive black/African American patients with type 2 diabetes mellitus. Curr Med Res Opin. 2018 Feb;34(2):361-367. doi: 10.1080/03007995.2017.1405800. Epub 2017 Nov 29. PMID 29139301

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this Phase 3b, multi-centre trial, a total of 719 patients were screened by 92 centres across the United States. The first centre was initiated on 25 Jul 2014. Of the 719 screened patients, 297 patients entered the placebo run-in phase of the trial and 166 were subsequently randomised to double-blind treatment
Pre-assignment Details: Empagliflozin was administered at a starting dose of 10 milligram (mg) once daily. At Week 4, patients were dose escalated to a dose of 25 mg once daily. These doses were selected based on the results from previous dose-finding studies
Groups:
- Placebo: Patients were orally administered Placebo matching empagliflozin 10 mg or 25 mg (1 tablet once daily, morning)
- Empagliflozin 10 Mg-25mg: Patients were orally administered Empagliflozin 10 mg or 25mg (1 tablet once daily, morning over a period of 24 weeks)
Period: Overall Study
Arm/Group | Placebo | Empagliflozin 10 Mg-25mg
Started | 83 | 83
Randomised Set (RS) (Randomised Patients screened for trial, regardless of whether any trial drug was taken.) | 79 (From started, 2 duplicate patients and 2 patients from one site were removed) | 82 (From started, 1 patient from one site was removed)
Treated Set (TS) (All patients in the RS who received at least one dose of trial medication.) | 77 (From RS, 1 duplicate patient and 1 non treated patient was removed) | 80 (From RS, 1 duplicate patient and 1 non treated patient was removed)
Completed | 68 | 68
Not Completed | 15 | 15
Not completed — Not Treated | 1 | 1
Not completed — Trial stopped, reason missing | 3 | 3
Not completed — Consent withdrawn | 8 | 8
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): All patients randomised, treated with at least one dose of trial drug, and with a baseline and at least one on-treatment glycated haemoglobin (HbA1c)value. The FAS was the basis for the primary efficacy analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Empagliflozin 10 Mg-25mg | Total
Number analyzed (Participants) | 72 | 78 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Full analysis set (FAS): All patients randomised, treated with at least one dose of trial drug, and with a baseline and at least one on-treatment HbA1c value. The FAS was the basis for the primary efficacy analysis.
  years | 57.2 (9.3) | 56.5 (9.3) | 56.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: FAS
  Participants
    Female | 36 | 35 | 71
    Male | 36 | 43 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: FAS
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 72 | 78 | 150
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: FAS
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 72 | 78 | 150
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Baseline hemoglobin A1c (HbA1c) [%] [Mean (Standard Deviation); unit: percentage of HbA1c] — Mean and standard deviation for Baseline HbA1c [%] is presented Population: FAS
  percentage of HbA1c | 8.51 (1.12) | 8.66 (0.92) | 8.59 (1.02)
Baseline estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m²] — Population: FAS
  mL/min/1.73m² | 91.49 (20.79) | 91.15 (18.95) | 91.31 (19.79)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycated Haemoglobin (HbA1c) (%) at 24 Weeks
Description: Change from baseline in HbA1c (%) at 24 weeks is presented. The term "baseline" refers to the last observation prior to randomisation of the patient.
  Means presented are the adjusted means. Restricted maximum likelihood (REML)-based mixed model repeated measures (MMRM) model is used in the statistical analysis.
Time Frame: baseline and 24 weeks
Population: Full analysis set (FAS) observed cases (OC); FAS: All patients randomised, treated with at least one dose of trial drug, and with a baseline and at least one on-treatment HbA1c value.
  Observed cases will set all values measured after antidiabetic rescue medication to missing
Measure: Mean (Standard Error); unit: percentage of glycated haemoglobin
Arm/Group | Placebo | Empagliflozin 10 Mg-25mg
Number analyzed (Participants) | 72 | 78
percentage of glycated haemoglobin | 0.07 (0.14) | -0.71 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 Mg-25mg; MMRM model : "HbA1c baseline," "treatment," "renal function," "pre-treatment with metformin," "visit," "visit by treatment interaction," and "HbA1c baseline by treatment interaction." "Treatment," "renal function," "pre-treatment with metformin," "visit," and "visit by treatment interaction" were fixed classification effects, and "HbA1c baseline" was a linear covariate. The interaction "visit by HbA1c baseline interaction" was based on the linear covariate "HbA1c baseline."; Test type: Superiority — A hierarchical multiple testing procedure was used to evaluate superiority of the primary endpoint; p = 0.0002, Mixed Models Analysis; Adjusted mean difference = -0.78, 95% CI 2-sided [-1.18 to -0.38], Standard Error of Mean 0.20 — Empagliflozin minus Placebo

2. Secondary Outcome: Change From Baseline in Mean 24-hour Ambulatory Systolic Blood Pressure (SBP) at Week 12
Description: Change from baseline in mean 24-hour ambulatory Systolic blood pressure SBP at Week 12 is presented. The term "baseline" refers to the last observation prior to randomisation of the patient.
  Means presented are the adjusted means. This is a key secondary endpoint
Time Frame: baseline and 12 weeks
Population: FAS LOCF-H; LOCF-H= Last observation carried forward without values following antidiabetic rescue medication and/or a change in antihypertensive therapy
Measure: Mean (Standard Error); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Empagliflozin 10 Mg-25mg
Number analyzed (Participants) | 72 | 78
millimeter of mercury (mmHg) | -0.90 (1.47) | -6.10 (1.41)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 Mg-25mg; change from baseline in mean 24-hour ambulatory SBP at 12 weeks of treatment was evaluated by using an Analysis of Covariance (ANCOVA) model. The respective model included treatment, renal function, pretreatment with metformin, continuous baseline HbA1c, and continuous baseline of the endpoint; Test type: Superiority — A hierarchical multiple testing procedure was used to evaluate superiority of the endpoint; p = 0.0117, ANCOVA; Adjusted mean difference = -5.21, 95% CI 2-sided [-9.24 to -1.18], Standard Error of Mean 2.04 — Empagliflozin minus Placebo

3. Secondary Outcome: Changes From Baseline in Trough Mean Ambulatory SBP at Week 12
Description: Changes from baseline in trough mean ambulatory SBP at Week 12 is presented. The term "baseline" refers to the last observation prior to randomisation of the patient.
  Means presented are the adjusted means. This is a key secondary endpoint
Time Frame: baseline and 12 weeks
Population: FAS LOCF-H
Measure: Mean (Standard Error); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Empagliflozin 10 Mg-25mg
Number analyzed (Participants) | 72 | 78
millimeter of mercury (mmHg) | -1.00 (1.89) | -6.99 (1.80)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 Mg-25mg; ANCOVA mode: The respective model included treatment, renal function, pretreatment with metformin, continuous baseline HbA1c, and continuous baseline of the endpoint; Test type: Superiority — A hierarchical multiple testing procedure was used to evaluate superiority of the endpoint; p = 0.0237, ANCOVA; Adjusted mean difference = -5.99, 95% CI 2-sided [-11.16 to -0.81], Standard Error of Mean 2.62 — Empagliflozin minus Placebo

4. Secondary Outcome: Change From Baseline in Body Weight at Week 24
Description: Changes from baseline in body weight at Week 24 is presented. The term "baseline" refers to the last observation prior to randomisation of the patient.
  Means presented are the adjusted means. This is a key secondary endpoint
Time Frame: baseline and 24 weeks
Population: FAS OC
Measure: Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Placebo | Empagliflozin 10 Mg-25mg
Number analyzed (Participants) | 72 | 78
kilogram (kg) | -0.98 (0.42) | -2.21 (0.41)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 Mg-25mg; MMRM models modelling the key secondary endpoint with continuous baseline HbA1c, continuous baseline key secondary endpoint, treatment, renal function, pretreatment with metformin, visit, visit by treatment interaction, visit by continuous baseline HbA1c interaction, visit by continuous baseline key secondary endpoint; Test type: Superiority — A hierarchical multiple testing procedure was used to evaluate superiority of the endpoint; p = 0.0382, Mixed Models Analysis; Adjusted mean difference = -1.23, 95% CI 2-sided [-2.39 to -0.07], Standard Error of Mean 0.59 — Empagliflozin minus Placebo

5. Secondary Outcome: Change From Baseline in Trough Seated SBP at Week 12
Description: Change from baseline in trough seated SBP (mmHg) at Week 12 is presented. The term "baseline" refers to the last observation prior to randomisation of the patient.
  Means presented are the adjusted means. This is a key secondary endpoint
Time Frame: baseline and 12 weeks
Population: FAS OC-H =FAS observed cases without values following a change in antihypertensive therapy (OC-H)
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Empagliflozin 10 Mg-25mg
Number analyzed (Participants) | 72 | 78
mmHg | -3.94 (1.82) | -7.97 (1.83)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 Mg-25mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — A hierarchical multiple testing procedure was used to evaluate superiority of the endpoint; p = 0.1215, Mixed Models Analysis; Adjusted mean difference = -4.04, 95% CI 2-sided [-9.16 to 1.09], Standard Error of Mean 2.59 — Empagliflozin minus Placebo

6. Secondary Outcome: Change From Baseline in Mean 24-hour Ambulatory SBP (mmHg) at Week 24
Description: Change from baseline in mean 24-hour ambulatory SBP (mmHg) at Week 24 is secondary endpoint. The term "baseline" refers to the last observation prior to randomisation of the patient.
  Means presented are the adjusted means.
Time Frame: baseline and 24 weeks
Population: FAS OC-H =FAS observed cases without values following a change in antihypertensive therapy (OC-H)
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Empagliflozin 10 Mg-25mg
Number analyzed (Participants) | 72 | 78
mmHg | -1.94 (1.94) | -10.33 (1.85)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 Mg-25mg; MMRM models modelling the secondary endpoint with continuous baseline HbA1c, continuous baseline secondary endpoint, treatment, renal function, pretreatment with metformin, visit, visit by treatment interaction, visit by continuous baseline HbA1c interaction, visit by continuous baseline secondary endpoint; Test type: Superiority; p = 0.0025, Mixed Models Analysis; Adjusted mean difference = -8.39, 95% CI 2-sided [-13.74 to -3.04], Standard Error of Mean 2.69 — Empagliflozin minus Placebo

7. Secondary Outcome: Change From Baseline in Mean 24-hour Ambulatory Diastolic Blood Pressure (DBP) at Week 12
Description: Change from baseline in mean 24-hour ambulatory DBP (mmHg) at Week 12. The term "baseline" refers to the last observation prior to randomisation of the patient.
  Means presented are the adjusted means.
Time Frame: baseline and 12 weeks
Population: FAS (LOCF-H)
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Empagliflozin 10 Mg-25mg
Number analyzed (Participants) | 72 | 78
mmHg | -0.37 (0.90) | -3.80 (0.86)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 Mg-25mg; The respective ANCOVA model includes treatment, renal function, pretreatment with metformin, continuous baseline HbA1c, and continuous baseline of the respective secondary endpoint; Test type: Superiority; p = 0.0069, ANCOVA; Adjusted mean difference = -3.43, 95% CI 2-sided [-5.90 to -0.96], Standard Error of Mean 1.25 — Empagliflozin minus Placebo

8. Secondary Outcome: Change From Baseline in Mean 24-hour Ambulatory DBP (mmHg) at Week 24
Description: Change from baseline in mean 24-hour ambulatory DBP (mmHg) at Week 24 is secondary endpoint. The term "baseline" refers to the last observation prior to randomisation of the patient.
  Means presented are the adjusted means.
Time Frame: baseline and 24 weeks
Population: FAS OC-H =FAS observed cases without values following a change in antihypertensive therapy (OC-H)
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Empagliflozin 10 Mg-25mg
Number analyzed (Participants) | 72 | 78
mmHg | -1.48 (1.24) | -6.38 (1.20)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 Mg-25mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0058, Mixed Models Analysis; Adjusted mean difference = -4.91, 95% CI 2-sided [-8.35 to -1.46], Standard Error of Mean 1.74 — Empagliflozin minus Placebo

9. Secondary Outcome: Change From Baseline in Trough Seated SBP (mmHg) at Week 24
Description: Change from baseline in trough seated SBP (mmHg) at Week 24 is secondary endpoint. The term "baseline" refers to the last observation prior to randomisation of the patient.
  Means presented are the adjusted means.
Time Frame: baseline and 24 weeks
Population: FAS OC-H =FAS observed cases without values following a change in antihypertensive therapy (OC-H)
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Empagliflozin 10 Mg-25mg
Number analyzed (Participants) | 72 | 78
mmHg | -2.83 (1.82) | -10.26 (1.70)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 Mg-25mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0036, Mixed Models Analysis; Adjusted mean difference = -7.43, 95% CI 2-sided [-12.37 to -2.48], Standard Error of Mean 2.50 — Empagliflozin minus Placebo

10. Secondary Outcome: Change From Baseline in Trough Seated DBP (mmHg) at Week 12
Description: Change from baseline in trough seated DBP (mmHg) at Week 12 is secondary endpoint. The term "baseline" refers to the last observation prior to randomisation of the patient.
  Means presented are the adjusted means.
Time Frame: baseline and 12 weeks
Population: FAS OC-H =FAS observed cases without values following a change in antihypertensive therapy (OC-H)
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Empagliflozin 10 Mg-25mg
Number analyzed (Participants) | 72 | 78
mmHg | -2.30 (1.09) | -4.14 (1.10)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 Mg-25mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.2402, Mixed Models Analysis; Adjusted mean difference = -1.84, 95% CI 2-sided [-4.93 to 1.25], Standard Error of Mean 1.56 — Empagliflozin minus Placebo

11. Secondary Outcome: Change From Baseline in Trough Seated DBP (mmHg) at Week 24
Description: Change from baseline in trough seated DBP (mmHg) at Week 24 is secondary endpoint. The term "baseline" refers to the last observation prior to randomisation of the patient.
  Means presented are the adjusted means.
Time Frame: baseline and 24 weeks
Population: FAS OC-H =FAS observed cases without values following a change in antihypertensive therapy (OC-H)
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Empagliflozin 10 Mg-25mg
Number analyzed (Participants) | 72 | 78
mmHg | -1.30 (1.09) | -5.55 (1.02)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 Mg-25mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0053, Mixed Models Analysis; Adjusted mean difference = -4.25, 95% CI 2-sided [-7.21 to -1.29], Standard Error of Mean 1.49 — Empagliflozin minus Placebo

ADVERSE EVENTS:
Time Frame: All adverse events occurring after the first dose of trial medication up to a period of 7 days after the last dose of trial medication (i.e. end of REP); up to 25 weeks
Description: All the safety analyses were based on treated set except the serious adverse event analysis. The two patients with multiple participation in the study (counted once as first randomized) and three patients excluded from one site were included back into treated set for the analysis of serious adverse event.
Arm/Group | Placebo | Empagliflozin 10 Mg-25mg
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/82
Serious Adverse Events (participants affected / at risk) | 4/80 | 3/82
Other Adverse Events (participants affected / at risk) | 8/77 | 12/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=80) | Empagliflozin 10 Mg-25mg (N=82)
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=77) | Empagliflozin 10 Mg-25mg (N=80)
Lipase increased (Investigations) | 3 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT02182830/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT02182830/SAP_001.pdf